CLINICAL TRIAL: NCT06449781
Title: 177Lu-PSMA as a Systemic Adjuvant Treatment in Patients With High- and Very High-risk Prostate Cancer After Radical Treatment Using Locoregional Teleradiotherapy and Hormone Therapy
Brief Title: 177Lu-PSMA as a Systemic Adjuvant Treatment in Patients With High and Very High Risk Prostate Cancer
Acronym: PSMA-ADJUVO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSMA-ADJUVO; Nr EU CT: 2023-504912-13-00 (Other: EMA)
Record Dates: First submitted 2023-12-06; First posted 2024-06-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium; Lutetium-177; Pluvicto

STUDY DESIGN:
Intervention Model Description: Open-label, two-arm, randomized study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): The intervention will consist of a single administration of 177Lu-PSMA with an activity of 7.4 GBq. Participants will also receive standard hormone therapy
  Interventions: Drug: Lutetium (177Lu) vipivotide tetraxetan
- Control (No Intervention): Participants will receive standard hormone therapy

INTERVENTIONS:
Drug: Lutetium (177Lu) vipivotide tetraxetan — The intervention will consist of a single administration of 7,4 GBq of lutetium (177Lu) vipivotide tetraxetan
  Other Names: Pluvicto
  Arms: Experimental

SUMMARY:
Single-center, non-commercial phase 2 clinical trial to evaluate 177Lu-PSMA as a systemic adjuvant treatment in patients with high and very high risk prostate cancer after radical treatment using locoregional teleradiotherapy and hormone therapy

DETAILED DESCRIPTION:
The intervention will consist of a single administration of 177Lu-PSMA in the research arm. Both the study and control groups will receive standard hormone therapy.

The study population includes 200 adult men with high-risk or very high-risk prostate cancer, with no signs of cancer dissemination in radiological examinations after completion of radiotherapy and continued hormone therapy

Participation time in the Study:

intervention phase - 1 day; observation phase - 5 years

ELIGIBILITY:
Inclusion Criteria:

* Giving a written informed consent
* Histopathologically confirmed high or very high risk prostate cancer
* Completion of radical locoregional treatment
* Completion of locoregional treatment within 3 months before inclusion to the study
* ECOG performance status 0 to 2
* Age over 18 years
* Within 28 days before entering the study, there were no signs of cancer dissemination documented in radiological tests
* Castrate testosterone level (testosteron < 50 ng/dL lub 1,7 nmol/L)
* Patients with adequate function of main organs:

  * bone marrow:

    * neutrophils > 1500x10^9/L;
    * thrombocytes > 100,000x10^9/L;
    * hemoglobin > 9 g/dL
  * liver:

    * bilirubin < 2xULN (upper limit of normal) in patients with Gilbert's syndrome < 5xULN;
    * aminotransferase < 3xULN
  * kidneys:

    * eGFR > 50 ml/min
    * albumin >2.5 mg/ml
* For men of reproductive age: the need to use double barrier contraception

Exclusion Criteria:

* The presence of distant metastases confirmed by radiological examination
* Absence of approval to use effective contraception method
* Absence of Patient's consent to participate in the Study
* Urinary tract obstruction or/and hydronephrosis.
* Concurrent anticancer treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness | 2 and 5 years after end of treatment
  Assessment of treatment failure - the assesment of biochemical progression ratio, defined as a rise of PSA by 2 ng/mL or more above the nadir, proven by a consecutive examination performed at least 4 weeks later

SECONDARY OUTCOMES:
Biochemical progression-free survival | During the intervention and follow up period (assessed up to 5 years)
  Comparative assessment of biochemical progression-free survival time defined as an increase in tPSA (prostate specific antigen) in the blood above the nadir (the lowest PSA value after completion of treatment) by 2 ng/mL or more, confirmed in the next test performed no earlier than after 4 weeks
Radiological progression-free survival | During the intervention and follow up period (assessed up to 5 years)
  Comparative assessment of radiological progression-free survival defined according to PCWG3 criteria
Time until the next therapeutic intervention | During the intervention and follow up period (assessed up to 5 years)
  Comparative assessment of the time until the next therapeutic intervention
Incidence of Treatment-Emergent Adverse Events according to CTCAE v 5.0 | During the intervention and follow up period (assessed up to 5 years)
  Comparative assessment of safety and tolerability of treatment according to CTCAE v 5.0
Quliaty of life | During the intervention and follow up period (assessed up to 5 years)
  Comparison of EORTC QLQ-PR25 quality of life indicators between study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch, Gliwice, Poland

IPD SHARING:
Plan to Share IPD: No